CLINICAL TRIAL: NCT01853345
Title: Individualized Cancer Therapy (iCAT) Recommendation for Patients With Recurrent, Refractory or High Risk Solid Tumors
Brief Title: iCAT for Recurrent/Refractory/HR Solid Tumors
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Katherine Janeway, MD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 11-406
Record Dates: First submitted 2013-04-25; First posted 2013-05-15 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Pediatric Solid Tumor; Sarcoma; Neuroblastoma; Wilms Tumor
Keywords: Refractory; Recurrent; High Risk
MeSH Terms: conditions — Sarcoma; Neuroblastoma; Wilms Tumor; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 99 Years
Biospecimen Retention: Samples With DNA — Blood samples, tumor samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Refractory/Recurrent/High Risk Solid Tumors

SUMMARY:
In this study tumor will be tested for cancer causing gene alterations such as mutations or copy number alterations. This is called tumor profiling. A panel of experts will review the tumor profiling results and determine whether there is a cancer-causing alteration present in the tumor. If there is, the experts will determine if there is a targeted drug available that could counteract this alteration. If there is an alteration identified and a targeted drug available the panel of experts will make an individualized treatment recommendation. The results of the tumor profiling and the individualized treatment recommendation can be shared with the primary oncologist.

DETAILED DESCRIPTION:
Some cancer-causing gene alterations (such as mutations or copy number alterations) are common or occur repeatedly in different types of cancers. For some of these alterations there are drugs, called targeted drugs that specifically counteract the alteration. In certain cancer types, these targeted drugs are very effective at fighting the cancer.

A tumor specimen that has been obtained previously or is planned to be obtained as part of clinical care will be used to perform tumor profiling. Additional procedures to obtain tumor will not be performed. An expert panel will review the results of the tumor profiling tests and determine whether a cancer-causing alteration is present and whether an individualized treatment recommendation can be made. If consent to sharing of the tumor profiling results and individualized treatment recommendation is provided then a study physician will discuss the profiling results and the individualized treatment recommendation with the primary oncologist. In addition, the primary oncologist will receive a letter detailing the tumor profiling results and the individualized treatment recommendation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent, refractory of high risk pediatric solid tumor (excluding brain tumor)
* Histologic proof of malignancy at the time of diagnosis or recurrence
* Sufficient tumor specimen available for profiling from diagnosis or recurrence, or surgery/biopsy planned for clinical care

Exclusion Criteria:

* Brain tumors

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with recurrent, refractory or high risk solid tumors
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2012-08; Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Frequency of a cancer causing actionable alteration and individualized treatment recommendation. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Janeway, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - University of California, San Francisco, San Francisco, California
  - Children's National Medical center, Washington D.C., District of Columbia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Columbia University, New York, New York

REFERENCES:
- [Derived] Harris MH, DuBois SG, Glade Bender JL, Kim A, Crompton BD, Parker E, Dumont IP, Hong AL, Guo D, Church A, Stegmaier K, Roberts CWM, Shusterman S, London WB, MacConaill LE, Lindeman NI, Diller L, Rodriguez-Galindo C, Janeway KA. Multicenter Feasibility Study of Tumor Molecular Profiling to Inform Therapeutic Decisions in Advanced Pediatric Solid Tumors: The Individualized Cancer Therapy (iCat) Study. JAMA Oncol. 2016 May 1;2(5):608-615. doi: 10.1001/jamaoncol.2015.5689. PMID 26822149